CLINICAL TRIAL: NCT04117191
Title: Exploring the Mechanisms of Indoxyl Sulfate Production by Oral Tryptophan Challenge Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Ting-Yun Lin, Nephrologist, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 08-P-055
Record Dates: First submitted 2019-09-29; First posted 2019-10-07 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Healthy; Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: All the participants would be introduced to receive 2g tryptophan loading for exploring serum and urine indoxyl sulfate concentration.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tryptophan loading (Experimental): All participants are introduced to receive tryptophan loading test.
  Interventions: Dietary Supplement: Doctor's Best L-Tryptophan

INTERVENTIONS:
Dietary Supplement: Doctor's Best L-Tryptophan — 2g tryptophan loading once

SUMMARY:
Cardiovascular disease (CVD) is prevalent in patients with chronic kidney disease (CKD) and is associated with extremely poor prognosis. Traditional risk factors for the general population, such as diabetes mellitus, high blood pressure, and dyslipidemia, are more common in patients with CKD but cannot fully explain the increased risk of this population. New evidence suggests that the uremic milieu itself plays a critical role in the development and progression of CVD. The gut microbiota is markedly altered in CKD, with overgrowth of bacteria that produce uremic toxins. Indoxyl sulfate (IS) is among the most representative gut-derived uremic toxins and has been most frequently implicated as a contributor to the pathogenesis of CVD in CKD. IS is converted from indole, a gut bacteria metabolite of dietary tryptophan, by two hepatic enzymes, CYP2E1 and SULT1A1. The majority of studies have assessed IS toxicity in cultured cells and animal models. However, human data have been conflicting and the benefit of using orally administered adsorbents to reduce IS levels in unselected CKD patients was not supported by results from the recent randomized controlled trials. IS levels may fluctuate widely from time to time with dietary intakes. The investigators hypothesize that a postprandial IS concentration may more reflect its toxicity than a single time point (fasting or predialysis IS) concentration measured in clinical studies. Therefore, the investigators plan to establish an oral tryptophan challenge test (OTCT) by using an oral loading of 2 gm tryptophan to simulate the postprandial increase of plasma IS. The investigators will recruit 60 healthy volunteers to undergo OTCT. A pharmacokinetic study of IS after the OTCT will be performed in 20 of them to verify and simplify the design of OTCT protocol. The results of OTCT will be integrated with whole metagenome analysis of fecal microbiota and genetic polymorphism analysis of CYP2E1 and SULT1A1 to explore the mechanisms of IS production. In addition to the known genes in microbe produces indoles, other supporting bacteria or genes will be examined by using metagenomic shotgun sequencing data.

ELIGIBILITY:
Inclusion Criteria:

* (1) age older than 20 years
* (2) no exposure to antibiotics or probiotics within the 3 months before entering the study.

Exclusion Criteria:

* (1) recent gastrointestinal discomfort (such as nausea, vomiting, abdominal pain, constipation, or diarrhea) or
* (2) a history of chronic diseases including diabetes mellites, hypertension, CVD, CKD, liver disease, malignancy, and autoimmune disease.
* (3) pregnancy or breast feeding
* (4) currently use of antipsychotics, Hypnotics, Demerol, Dextromethorphan, tramadol, pentazocine

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Indoxyl sulfate | the area under curve of serum and urine indoxyl sulfate within 72 hours
  serum and urine indoxyl sulfate concentration measurement

SECONDARY OUTCOMES:
Indole-3-acetic acid | the area under curve of serum and urine Indole-3-acetic acid within 72 hours
  serum and urine Indole-3-acetic acid concentration measurement

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Yun Lin, MD., Principal Investigator — Taichung Tzu Chi Hospital
Locations (1):
- Taipei Tzu Chi Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No